CLINICAL TRIAL: NCT01970488
Title: A Phase 3, Multicenter, Randomized, Double-blind Study Evaluating the Efficacy and Safety of ABP 501 Compared With Adalimumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Compare Efficacy and Safety of ABP 501 and Adalimumab (HUMIRA®) in Adults With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120263; 2013-000537-12 (EudraCT Number)
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; ABP 501

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 501 (Experimental): Participants received 80 mg ABP 501 subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter until week 16.
  Participants with a PASI 50 response at week 16 continued to receive 40 mg APB 501 until week 48.
  Interventions: Biological: ABP 501
- Adalimumab (Active Comparator): Participants received 80 mg adalimumab subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter until week 16.
  At week 16 participants with a PASI 50 response were re-randomized to treatment with adalimumab or were transitioned to ABP 501 until week 48.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Administered by subcutaneous injection
  Other Names: HUMIRA®
  Arms: Adalimumab
Biological: ABP 501 — Administered by subcutaneous injection
  Other Names: Adalimumab-atto; AMJEVITA™
  Arms: ABP 501

SUMMARY:
The purpose of this research study is to compare the efficacy and safety of ABP 501 and adalimumab (HUMIRA®) in adults with plaque psoriasis.

ELIGIBILITY:
Inclusion criteria:

1. Men or women ≥ 18 and ≤ 75 years of age at time of screening
2. Stable moderate to severe plaque psoriasis for at least 6 months before baseline
3. Moderate to severe psoriasis defined at screening and baseline by:

   Body surface area (BSA) affected by plaque psoriasis of 10% or greater, and PASI score of 12 or greater, and static physician's global assessment score of 3 or greater
4. No known history of active tuberculosis
5. Subject is a candidate for systemic therapy or phototherapy procedures
6. Previous failure, inadequate response, intolerance, or contraindication to at least 1 conventional anti-psoriatic systemic therapy

Exclusion Criteria:

1. Forms of psoriasis or other skin conditions at the time of the screening visit (eg, eczema)
2. Ongoing use of prohibited treatments
3. Prior use of 2 or more biologics for treatment of psoriasis
4. Previous receipt of adalimumab or a biosimilar of adalimumab

Other Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2014-08-14 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- Research Site, Saint Leonards, New South Wales, Australia
- Research Site, St. John's, Newfoundland and Labrador, Canada
- Research Site, Nyíregyháza, Szabolcs-Szatmár-Bereg, Hungary

REFERENCES:
- [Derived] Papp K, Bachelez H, Costanzo A, Foley P, Gooderham M, Kaur P, Philipp S, Spelman L, Zhang N, Strober B. Clinical similarity of the biosimilar ABP 501 compared with adalimumab after single transition: long-term results from a randomized controlled, double-blind, 52-week, phase III trial in patients with moderate-to-severe plaque psoriasis. Br J Dermatol. 2017 Dec;177(6):1562-1574. doi: 10.1111/bjd.15857. Epub 2017 Dec 1. PMID 28755394
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 49 centers in 6 countries (Australia, Canada, France, Germany, Hungary, and Poland).
  Participants were randomized in a 1:1 ratio to receive ABP 501 or adalimumab.
Pre-assignment Details: Randomization was stratified based on prior biologic use for psoriasis and geographic region. At week 16 participants with a PASI 50 response (≥ 50% improvement in Psoriasis Area and Severity Index score) continued on study; those initially randomized to adalimumab were re-randomized to receive either ABP 501 or adalimumab.
Groups:
- Part 1: ABP 501: Participants received 80 mg ABP 501 subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter for 16 weeks.
- Part 1: Adalimumab: Participants received 80 mg adalimumab subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter for 16 weeks.
- Part 2: ABP 501/ABP 501: Participants who received ABP 501 in Part 1 with a PASI 50 response at week 16 continued to receive 40 mg ABP 501 every 2 weeks until week 48.
- Part 2: Adalimumab/Adalimumab: Participants who received adalimumab in Part 1 with a PASI 50 response at week 16 continued to receive 40 mg adalimumab every 2 weeks until week 48.
- Part 2: Adalimumab/ABP 501: Participants who received adalimumab in Part 1 with a PASI 50 response at week 16 were transitioned to receive 40 mg ABP 501 every 2 weeks until week 48.
Period: Part 1: Through Week 16
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Started | 175 | 175 | 0 | 0 | 0
Received Treatment | 174 | 173 | 0 | 0 | 0
Completed | 164 | 162 | 0 | 0 | 0
Not Completed | 11 | 13 | 0 | 0 | 0
Not completed — Protocol-specified Criteria | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0
Period: Part 2: Post Week 16
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Started | 0 | 0 | 152 (Only participants who completed week 16 and with a PASI 50 response continued in Part 2) | 79 (Only participants who completed week 16 and with a PASI 50 response continued in Part 2) | 77 (Only participants who completed week 16 and with a PASI 50 response continued in Part 2)
Completed | 0 | 0 | 135 | 71 | 69
Not Completed | 0 | 0 | 17 | 8 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 5 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Total
Number analyzed (Participants) | 175 | 175 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.95) | 44.0 (13.68) | 44.6 (13.31)
Age, Customized [Number; unit: participants]
  < 65 years | 164 | 163 | 327
  ≥ 65 years | 11 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 59 | 122
  Male | 112 | 116 | 228
Race/Ethnicity, Customized [Number; unit: participants]
  White | 167 | 157 | 324
  Black or African American | 0 | 2 | 2
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Mixed Race | 0 | 1 | 1
  Other | 1 | 3 | 4
  Unknown | 2 | 3 | 5
Prior Biological Use for Psoriasis [Number; unit: participants]
  Yes | 33 | 30 | 63
  No | 142 | 145 | 287
Geographic Region [Number; unit: participants]
  Eastern Europe | 71 | 70 | 141
  Western Europe | 43 | 43 | 86
  Other | 61 | 62 | 123
Static Physician's Global Assessment (sPGA) [Number; unit: participants] — The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema).
  participants
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 106 | 102 | 208
    Severe | 61 | 61 | 122
    Very Severe | 7 | 10 | 17
    Missing | 1 | 2 | 3
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease.
  Data are reported for 174 and 173 participants in each reporting group respectively.
  units on a scale | 19.68 (8.100) | 20.48 (7.880) | 20.08 (7.990)
Body Surface Area (BSA) Affected by Psoriasis [Mean (Standard Deviation); unit: percentage of BSA] — Data are reported for 174 and 173 participants in each reporting group respectively.
  percentage of BSA | 25.3 (15.02) | 28.5 (16.82) | 26.9 (16.00)

OUTCOME MEASURES:

1. Primary Outcome: Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) at Week 16
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline was calculated as (value at baseline - value at post-baseline visit) × 100 / (value at baseline).
Time Frame: Baseline and Week 16
Population: This analysis was performed using the full analysis set which includes all participants initially randomized in the study. Last observation carried forward (LOCF) imputation was used for participants with at least one post-baseline value.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percent change | 80.91 (24.237) | 83.06 (25.195)
Statistical Analysis 1: Comparison: Part 1: ABP 501 vs Part 1: Adalimumab; Test type: Non-Inferiority or Equivalence — Clinical equivalence was evaluated by comparing the 2-sided 95% confidence interval (CI) of the difference of PASI percent improvement from baseline to Week 16 between ABP 501 and adalimumab with an equivalence margin of ± 15; Least Squares (LS) Mean Difference = -2.18, 95% CI 2-sided [-7.39 to 3.02]

2. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Week 16
Description: A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Week 16
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percentage of participants | 74.4 | 82.7

3. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Week 32
Description: as for outcome 2
Time Frame: Baseline and week 32
Population: This analysis was performed in the re-randomized analysis set which includes all participants who were re-randomized at Week 16 in the study. Only participants with available data at week 32 are included.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percentage of participants | 82.5 | 84.7 | 84.5

4. Secondary Outcome: Percentage of Participants With a PASI 75 Response at Week 50
Description: as for outcome 2
Time Frame: Baseline and week 50
Population: This analysis was performed in the re-randomized analysis set which includes all participants who were re-randomized at Week 16 in the study. Only participants with available data at week 50 are included.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percentage of participants | 85.1 | 87.1 | 81.2

5. Secondary Outcome: Percent Improvement From Baseline in PASI at Week 32
Description: The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline is calculated as (value at baseline - value at post-baseline visit) × 100 / (value at baseline).
Time Frame: Baseline and week 32
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percent change | 87.62 (18.387) | 88.16 (18.181) | 86.98 (16.637)

6. Secondary Outcome: Percent Improvement From Baseline in PASI at Week 50
Description: as for outcome 5
Time Frame: Baseline and week 50
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percent change | 87.16 (19.559) | 88.11 (20.957) | 85.82 (21.864)

7. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) Response at Week 16
Description: The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response is defined as a sPGA value of clear (score 0) or almost clear (score 1).
Time Frame: Week 16
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percentage of participants | 58.7 | 65.3

8. Secondary Outcome: Percentage of Participants With a sPGA Response at Week 32
Description: as for outcome 7
Time Frame: Week 32
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percentage of participants | 66.4 (18.387) | 72.2 (18.181) | 70.4 (16.637)

9. Secondary Outcome: Percentage of Participants With a sPGA Response at Week 50
Description: as for outcome 7
Time Frame: Week 50
Population: This analysis was performed in the re-randomized analysis set with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percentage of participants | 68.7 | 74.3 | 69.6

10. Secondary Outcome: Change From Baseline in the Percentage of Body Surface Area (BSA) Involved With Psoriasis at Week 16
Description: A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The percent of BSA affected was estimated by assuming that the subject's palm, excluding the fingers and thumb, represented roughly 1% of the body's surface.
  Change from baseline is calculated as (value at post-baseline visit - value at baseline).
  A decrease from baseline (negative value) indicates improvement.
Time Frame: Baseline and Week 16
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percentage of BSA | -18.0 (13.57) | -22.1 (17.11)

11. Secondary Outcome: Change From Baseline in the Percentage of BSA Involved With Psoriasis at Week 32
Description: as for outcome 10
Time Frame: Baseline and week 32
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percentage of BSA | -20.6 (13.87) | -25.3 (15.94) | -23.8 (16.17)

12. Secondary Outcome: Change From Baseline in the Percentage of BSA Involved With Psoriasis at Week 50
Description: as for outcome 10
Time Frame: Baseline and week 50
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percentage of BSA | -20.7 (13.58) | -25.5 (16.14) | -25.1 (17.43)

13. Secondary Outcome: Number of Participants With Adverse Events
Description: The Investigator assessed whether each adverse event (AE) was possibly related to the investigational product. AEs were graded for severity according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03.
  A serious AE is defined as an AE that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. Results are reported from Day 1 to week 16 for the Part 1 ABP 501 and Adalimumab groups, and from post week 16 to the end of study (week 52) for the Part 2 ABP 501/ABP 501, Adalimumab/Adalimumab and Adalimumab/ABP 501 groups.
Time Frame: From first dose of study drug until 28 days after the last dose. Treatment was for 16 weeks in Part 1 and 32 weeks in Part 2.
Population: The safety analysis set includes all randomized participants who received at least 1 dose of study drug, based on actual treatment received.
Measure: Number; unit: participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 174 | 173 | 152 | 79 | 77
participants
  Any adverse event (AE) | 117 | 110 | 108 | 52 | 54
  Grade ≥ 3 adverse event | 8 | 5 | 7 | 2 | 3
  Treatment-related adverse event (TRAE) | 43 | 43 | 28 | 18 | 20
  Grade ≥ 3 treatment-related adverse event | 4 | 2 | 3 | 1 | 1
  Serious adverse event (SAE) | 6 | 5 | 4 | 4 | 4
  Treatment-related serious adverse event | 4 | 0 | 2 | 1 | 1
  AE leading to discontinuation of study drug | 7 | 5 | 7 | 1 | 3
  TRAE leading to discontinuation of study drug | 4 | 3 | 3 | 1 | 2
  AE leading to discontinuation from study | 7 | 5 | 4 | 1 | 2
  TRAE leading to discontinuation from study | 4 | 3 | 2 | 1 | 1

14. Secondary Outcome: Percentage of Participants Developing Antibodies to ABP 501 or Adalimumab
Description: Two validated assays were used to detect the presence of anti-drug antibodies. Samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect anti-drug antibodies (ADA) against ABP 501 and adalimumab (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a non-cell based bioassay to determine neutralizing activity against ABP 501 or adalimumab (Neutralizing Antibody Assay).
  Developing antibody incidence is defined as a negative or no antibody result at baseline and a positive antibody result at a post-baseline time point.
Time Frame: For 16 weeks in Part 1 and for 52 weeks for participants who were re-randomized in Part 2.
Population: Results are reported for the anti-drug antibody analysis set (defined as the subset of participants in the Safety Analysis Set who had at least 1 evaluable antibody test) from Baseline to Week 16 for all randomized participants, and from baseline to Week 52 for participants who were re-randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 174 | 173 | 152 | 79 | 77
percentage of participants
  Binding Antibody Positive | 55.2 | 63.6 | 68.4 | 74.7 | 72.7
  Neutralizing Antibody Positive | 9.8 | 13.9 | 13.8 | 20.3 | 24.7

15. Post Hoc Outcome: Percentage of Participants With a PASI 90 Response at Week 16
Description: A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Week 16
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percentage of participants | 47.1 | 47.4

16. Post Hoc Outcome: Percentage of Participants With a PASI 90 Response at Week 32
Description: as for outcome 15
Time Frame: Baseline and Week 32
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percentage of participants | 62.2 (18.387) | 65.3 (18.181) | 57.7 (16.637)

17. Post Hoc Outcome: Percentage of Participants With a PASI 90 Response at Week 50
Description: as for outcome 15
Time Frame: Baseline and Week 50
Population: This analysis was performed in the re-randomized analysis set with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percentage of participants | 59.0 | 64.3 | 66.7

18. Post Hoc Outcome: Percentage of Participants With a PASI 100 Response at Week 16
Description: A PASI 100 response is a 100% improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Time Frame: Baseline and Week 16
Population: Full analysis set; LOCF imputation was used for participants with at least 1 postbaseline value.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab
Number analyzed (Participants) | 172 | 173
percentage of participants | 16.9 | 19.7

19. Post Hoc Outcome: Percentage of Participants With a PASI 100 Response at Week 32
Description: as for outcome 18
Time Frame: Baseline and Week 32
Population: This analysis was performed in the re-randomized analysis set with available data
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 143 | 72 | 71
percentage of participants | 32.9 (18.387) | 33.3 (18.181) | 25.4 (16.637)

20. Post Hoc Outcome: Percentage of Participants With a PASI 100 Response at Week 50
Description: as for outcome 18
Time Frame: Baseline and Week 50
Population: This analysis was performed in the re-randomized analysis set with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Number analyzed (Participants) | 134 | 70 | 69
percentage of participants | 32.8 | 35.7 | 34.8

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 28 days after the last dose. Treatment was for 16 weeks in Part 1 and 32 weeks in Part 2.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Part 1: ABP 501 | Part 1: Adalimumab | Part 2: ABP 501/ABP 501 | Part 2: Adalimumab/Adalimumab | Part 2: Adalimumab/ABP 501
Serious Adverse Events (participants affected / at risk) | 6/174 | 5/173 | 4/152 | 4/79 | 4/77
Other Adverse Events (participants affected / at risk) | 50/174 | 60/173 | 48/152 | 31/79 | 34/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: ABP 501 (N=174) | Part 1: Adalimumab (N=173) | Part 2: ABP 501/ABP 501 (N=152) | Part 2: Adalimumab/Adalimumab (N=79) | Part 2: Adalimumab/ABP 501 (N=77)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: ABP 501 (N=174) | Part 1: Adalimumab (N=173) | Part 2: ABP 501/ABP 501 (N=152) | Part 2: Adalimumab/Adalimumab (N=79) | Part 2: Adalimumab/ABP 501 (N=77)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 4 | 8
Nasopharyngitis (Infections and infestations) | 25 | 27 | 25 | 14 | 18
Upper respiratory tract infection (Infections and infestations) | 9 | 9 | 9 | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 4 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 5 | 5 | 1
Headache (Nervous system disorders) | 12 | 18 | 5 | 8 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 2 | 10 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.